CLINICAL TRIAL: NCT00407745
Title: A 17-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Trial Of Pregabalin For The Treatment Of Chronic Central Neuropathic Pain After Spinal Cord Injury
Brief Title: A 17-Week Trial To Assess Pregabalin For The Treatment Of Nerve Pain Due To Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081107
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2012-02

CONDITIONS: Neuralgia; Spinal Cord Injuries
Keywords: Pain; central neuropathic pain
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- matched placebo (Placebo Comparator)
  Interventions: Drug: placebo
- pregabalin (Experimental): flexible dosing over 4 weeks followed by 12 weeks maintenance and one week taper period
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: placebo — Placebo
  Arms: matched placebo
Drug: pregabalin — Pregabalin capsules taken twice daily up to 17 weeks (150-600 mg/day)
  Other Names: Lyrica
  Arms: pregabalin

SUMMARY:
The purpose of this study is to evaluate if pregabalin relieves nerve pain associated with spinal cord injury compared to placebo (pill that contains no active medicine). This study will also evaluate the safety of pregabalin in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with nerve pain after Spinal cord injury (traumatic, diving, ischemic and after removal of benign tumors (except meningioma and fibromas)
* Pain has to be chronic(continuous for at least 3 months or intermittent for at least 6 months
* Pain score at least 4 in 4 of 7 days prior to receive treatment.

Exclusion Criteria:

* Pregabalin use in the last 60 days, prior intolerance to pregabalin
* Creatinine clearance <60 mL/min.
* White blood cell count <2500/mm3; neutrophil count <1500/mm3; platelet count <100 x 103/ mm3.
* Abuse of drugs or alcohol
* Unstable medial conditions
* Clinically significant abnormal electrocardiogram (ECG).
* Presence of severe pain associated with conditions other than spinal cord injury that could confound the assessment or self-evaluation of pain due to spinal cord injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (18):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Napa, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, White Plains, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bellevue, Ohio
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Charleston, West Virginia
- Pfizer Investigational Site, Viña del Mar, Región de Valparaíso, Chile
- China (3):
  - Pfizer Investigational Site, Beijing, Beijing Municipality
  - Pfizer Investigational Site, Chengdu, Sichuan
  - Pfizer Investigational Site, Beijing
- Pfizer Investigational Site, Medellín, Antioquia, Colombia
- Czechia (3):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Liberec
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Hong Kong, Hong Kong
- India (5):
  - Pfizer Investigational Site, Secunderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
  - Pfizer Investigational Site, New Delhi
- Japan (24):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Daisen, Akita
  - Pfizer Investigational Site, Iizuka, Fukuoka
  - Pfizer Investigational Site, Fukuyama, Hiroshima
  - Pfizer Investigational Site, Bibai, Hokkaido
  - Pfizer Investigational Site, Hakodate, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Sasima-gun, Ibaraki
  - Pfizer Investigational Site, Kawasaki, Kanagawa
  - Pfizer Investigational Site, Kikuchi-gun, Kumamoto
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Kashiwazaki, Niigata
  - Pfizer Investigational Site, Beppu, Oita Prefecture
  - Pfizer Investigational Site, Hanyū, Saitama
  - Pfizer Investigational Site, Kitamoto, Saitama
  - Pfizer Investigational Site, Hamamatsu, Shizuoka
  - Pfizer Investigational Site, Kanuma, Tochigi
  - Pfizer Investigational Site, Kotoku, Tokyo
  - Pfizer Investigational Site, Musashimurayama-shi, Tokyo
  - Pfizer Investigational Site, Higashiokitama-gun, Yamagata
  - Pfizer Investigational Site, Chiba
  - Pfizer Investigational Site, Tokushima
  - Pfizer Investigational Site, Yamagata
- Philippines (4):
  - Pfizer Investigational Site, España, Manila
  - Pfizer Investigational Site, Cebu City
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg

REFERENCES:
- [Derived] Schug SA, Parsons B, Almas M, Whalen E. Effect of Concomitant Pain Medications on Response to Pregabalin in Patients with Postherpetic Neuralgia or Spinal Cord Injury-Related Neuropathic Pain. Pain Physician. 2017 Jan-Feb;20(1):E53-E63. PMID 28072797
- [Derived] Markman JD, Jensen TS, Semel D, Li C, Parsons B, Behar R, Sadosky AB. Effects of Pregabalin in Patients with Neuropathic Pain Previously Treated with Gabapentin: A Pooled Analysis of Parallel-Group, Randomized, Placebo-controlled Clinical Trials. Pain Pract. 2017 Jul;17(6):718-728. doi: 10.1111/papr.12516. Epub 2016 Dec 1. PMID 27611736
- [Derived] Cardenas DD, Nieshoff EC, Suda K, Goto S, Sanin L, Kaneko T, Sporn J, Parsons B, Soulsby M, Yang R, Whalen E, Scavone JM, Suzuki MM, Knapp LE. A randomized trial of pregabalin in patients with neuropathic pain due to spinal cord injury. Neurology. 2013 Feb 5;80(6):533-9. doi: 10.1212/WNL.0b013e318281546b. Epub 2013 Jan 23. PMID 23345639
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081107&StudyName=A%2017-Week%20Trial%20To%20Assess%20Pregabalin%20For%20The%20Treatment%20Of%20Nerve%20Pain%20Due%20To%20Spinal%20Cord%20Injury

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was randomized after the first dose of study drug was taken; the participant was randomized to placebo, but the actual drug taken was pregabalin. This partcipant was included in the placebo group for all baseline characteristics and efficacy outcome measures; and in the pregabalin group for overall study and adverse events reporting.
Groups:
- Pregabalin: Pregabalin 75 milligram (mg) capsule administered by mouth (PO) twice daily (BID) for 7 days. On Day 8, dose may have been maintained at 150 mg per day or increased to 300 mg per day. Each week thereafter, including at Visit 4, a dose increase or decrease may have occurred depending on clinical judgement on adequate pain relief and tolerability. Following the end of adjustment phase, at Visit 4, participants were at their optimized dose (150 mg per day, 300 mg per day, 450 mg per day, or 600 mg per day). Participants remained at this maintenance dose throughout the next 12 weeks of the study.
- Placebo: Placebo matching study treatment.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 112 | 108
Treated | 112 | 107
Completed | 93 | 91
Not Completed | 19 | 17
Not completed — Lack of Efficacy | 1 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 5 | 3
Not completed — Adverse Event | 8 | 8
Not completed — Other | 2 | 0
Not completed — Randomized, unknown if treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 111 | 108 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] — 1 participant was randomized to placebo, but the actual drug taken was pregabalin. This subject was included in the placebo group for all baseline measures.
  years | 46.1 (12.7) | 45.6 (13.8) | 45.9 (13.3)
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 52 | 53 | 105
  Between 45 and 64 years | 50 | 45 | 95
  >= 65 years | 9 | 10 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 16 | 43
  Male | 84 | 92 | 176

OUTCOME MEASURES:

1. Primary Outcome: Duration Adjusted Average Change (DAAC) of Mean Pain Score
Description: DAAC was derived from participant's daily pain diary, where pain was measured on an 11-point Numerical Rating Scale (NRS-Pain)ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). The DAAC was calculated as the mean of all daily pain diary rating post baseline minus the baseline score then multiplied by the proportion of the planned study duration completed by the participant.
Time Frame: Baseline, Week 16
Population: mITT: all randomized participants who received at least one dose of study medication except the 8 participants who were randomized before protocol amendment 2.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale | -1.66 (0.157) | -1.07 (0.149)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis - the mean DAAC for the pregabalin group is equal to the mean DAAC for the placebo group; Alternative hypothesis - the mean DAAC for the placebo group differs from the mean DAAC for the pregabalin group. ANCOVA model included baseline severity of pain and Baseline Pain Catastrophizing Scale (PCS) Total Score as covariates and pooled center and treatment as fixed (class) cofactors; Test type: Superiority or Other; p = 0.0032, ANCOVA — Significance was declared if the 2-tailed test for the difference between treatment groups was significant at the 0.05 level; LS Mean Difference = -0.59, 95% CI 2-sided [-0.98 to -0.20], Standard Error of Mean 0.198

2. Secondary Outcome: Change From Baseline in Weekly Mean Pain Score
Description: Mean weekly score was calculated as the average of the available daily diary pain score values for the week. Pain score was measured on an 11-point numeric rating scale (NRS): 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 16
Population: mITT; modified baseline observation carried forward (mBOCF) imputation: mBOCF mean pain score was defined as the baseline mean pain score for participants who discontinued double-blind treatment due to adverse event or who had no postbaseline observations and as the last observation carried forward (LOCF) mean pain score for all other participants.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline | 6.5 (1.45) | 6.5 (1.41)
  Change from baseline at endpoint | -1.9 (1.91) | -1.2 (1.78)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.0066, ANCOVA — Serial gate-keeping multiple testing procedure was used. If primary comparison for DAAC was significant, then variables were assessed in a hierarchical manner. Significance was declared if unadjusted p-value was significant at 0.05 level (<=0.05); ANCOVA model included baseline severity (pain) and baseline PCS as covariates and effects for treatment and pooled center as fixed (class) cofactors; LS Mean Difference = -0.70, 95% CI 2-sided [-1.20 to -0.20], Standard Error of Mean 0.255

3. Secondary Outcome: Number of Participants With >=30% Reduction in Weekly Mean Pain Score From Baseline
Description: as for outcome 2
Time Frame: Baseline, Week 16
Population: mITT; LOCF: LOCF Endpoint corresponded to the last 7 days of diary data up to and including Week 16 and applied if the Week 16 assessment was missing; (N) = number of participants that can be analyzed for the endpoint.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 105
participants | 48 | 33
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis - The rate of responder for the pregabain group was equal to the rate of responder for the placebo group; Alternative hypothesis - The rate of responder for the pregabain group was not equal to the rate of responder for the placebo group; Test type: Superiority or Other; p = 0.0390, Regression, Logistic — Serial gate-keeping multiple testing was used. If primary comparison for DAAC was significant, then variables were assessed in hierarchical manner. Significance was declared if unadjusted p-value at 0.05 level and preceding tests were significant; Logistic regression model used terms for baseline pain score and baseline PCS total score as covariate, and pooled center and treatment as cofactor; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.032 to 3.328]

4. Secondary Outcome: Number of Participants With Categorical Scores on the Patient Global Impression of Change (PGIC) (Full Scale)
Description: The PGIC is a participant-rated instrument measuring change in the participant's overall status on a 7-point scale: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (N) = number of participants with data available for analysis
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 100 | 99
participants
  1-Very much improved | 7 | 2
  2-Much improved | 33 | 25
  3-Minimally improved | 38 | 24
  4-No change | 19 | 40
  5-Minimally worse | 2 | 5
  6-Much worse | 0 | 3
  7-Very much worse | 1 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis - The raw mean score for the pregabain group was equal to the raw mean score for the placebo group; Alternative hypothesis - The raw mean score for the pregabain group was not equal to the raw mean score for the placebo group; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Modified ridit transformation with the Cochran-Mantel- Haenszel test was used with adjusting for pooled center

5. Secondary Outcome: Change From Baseline in Weekly Mean Sleep Interference Score
Description: Pain-related sleep interference was assessed on an 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]).
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 105, 105) | 4.9 (2.48) | 5.2 (2.24)
  Change from baseline at endpoint (n = 105, 104) | -2.0 (2.35) | -1.0 (1.77)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; ANCOVA model included baseline sleep interference score as a covariate and pooled center and treatment as fixed (class) cofactors; LS Mean Difference = -1.08, 95% CI 2-sided [-1.60 to -0.56], Standard Error of Mean 0.265

6. Secondary Outcome: Change From Baseline in Weekly Mean Pain Score by Week
Description: as for outcome 2
Time Frame: Baseline, Week 1 through16
Population: ITT population: defined as all randomized participants who took at least one dose of study medication. (This population included the 8 participants who were randomized before the protocol amendment 2). (n) = number of participants with data for analysis.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 108
score on scale
  Baseline (n = 111, 108) | 6.44 (1.44) | 6.51 (1.40)
  Change at Week 1 (n = 111, 107) | -0.85 (1.04) | -0.38 (0.89)
  Change at Week 2 (n = 110, 105) | -1.26 (1.21) | -0.62 (1.30)
  Change at Week 3 (n = 107, 105) | -1.35 (1.35) | -0.86 (1.35)
  Change at Week 4 (n = 107, 103) | -1.64 (1.61) | -1.03 (1.53)
  Change at Week 5 (n = 105, 101) | -1.87 (1.73) | -1.07 (1.50)
  Change at Week 6 (n = 105, 99) | -1.89 (1.90) | -1.22 (1.72)
  Change at Week 7 (n = 103, 98) | -2.02 (1.86) | -1.34 (1.75)
  Change at Week 8 (n = 101, 97) | -1.96 (1.82) | -1.32 (1.82)
  Change at Week 9 (n = 98, 97) | -1.99 (1.81) | -1.37 (1.75)
  Change at Week 10 (n = 97, 91) | -2.03 (1.75) | -1.32 (1.81)
  Change at Week 11 (n = 96, 90) | -2.04 (1.82) | -1.43 (1.84)
  Change at Week 12 (n = 96, 91) | -1.90 (1.83) | -1.44 (1.93)
  Change at Week 13 (n = 93, 91) | -2.02 (1.76) | -1.39 (1.92)
  Change at Week 14 (n = 93, 92) | -2.00 (1.76) | -1.34 (1.89)
  Change at Week 15 (n = 93, 92) | -2.09 (1.80) | -1.41 (1.85)
  Change at Week 16 (n = 89, 90) | -2.17 (1.78) | -1.36 (1.87)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0295, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.49, 95% CI 2-sided [-0.94 to -0.05], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0033, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.67, 95% CI 2-sided [-1.11 to -0.22], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0185, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.54, 95% CI 2-sided [-0.98 to -0.09], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0040, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.66, 95% CI 2-sided [-1.10 to -0.21], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.81, 95% CI 2-sided [-1.26 to -0.36], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.72, 95% CI 2-sided [-1.17 to -0.27], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 7 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0027, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.69, 95% CI 2-sided [-1.14 to -0.24], Standard Error of Mean 0.23
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.66, 95% CI 2-sided [-1.11 to -0.21], Standard Error of Mean 0.23
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Week 9 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0058, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.64, 95% CI 2-sided [-1.09 to -0.18], Standard Error of Mean 0.23
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Week 10 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.69, 95% CI 2-sided [-1.14 to -0.23], Standard Error of Mean 0.23
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Week 11 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.62, 95% CI 2-sided [-1.08 to -0.17], Standard Error of Mean 0.23
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Week 12 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0328, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.50, 95% CI 2-sided [-0.95 to -0.04], Standard Error of Mean 0.23
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Week 13 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0150, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.57, 95% CI 2-sided [-1.02 to -0.11], Standard Error of Mean 0.23
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Week 14 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0048, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.66, 95% CI 2-sided [-1.11 to -0.20], Standard Error of Mean 0.23
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Week 15 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.69, 95% CI 2-sided [-1.15 to -0.24], Standard Error of Mean 0.23
Statistical Analysis 16: Comparison: Pregabalin vs Placebo; Week 16 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, study center, time (week), baseline pain score, baseline PCS total score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS Mean Difference = -0.76, 95% CI 2-sided [-1.22 to -0.30], Standard Error of Mean 0.23

7. Secondary Outcome: Number of Participants With >=50% Reduction in Weekly Mean Pain Score From Baseline
Description: as for outcome 2
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (N) = number of participants with data available for analysis
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 105
participants | 31 | 16
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0256, Regression, Logistic — Significance was declared if p-value <=0.05; Logistic regression used terms for treatment, baseline pain score as covariate, baseline PCS total score, and pooled center as cofactor; Odds Ratio (OR) = 2.24, 95% CI 2-sided [1.103 to 4.546]

8. Other Pre Specified Outcome: Change From Baseline in Weekly Mean Sleep Interference Score by Week
Description: Pain related sleep interference was assessed on an 11 point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]).
Time Frame: Baseline, Week 1 through 16
Population: ITT; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 108
score on scale
  Baseline (n = 111, 107) | 4.86 (2.46) | 5.18 (2.23)
  Change at Week 1 (n = 111, 106) | -0.96 (1.45) | -0.26 (0.85)
  Change at Week 2 (n = 110, 104) | -1.29 (1.63) | -0.49 (1.17)
  Change at Week 3 (n = 107, 104) | -1.36 (1.68) | -0.61 (1.27)
  Change at Week 4 (n = 107, 102) | -1.59 (1.85) | -0.90 (1.45)
  Change at Week 5 (n = 105, 100) | -1.81 (2.05) | -0.91 (1.38)
  Change at Week 6 (n = 105, 98) | -1.86 (2.14) | -0.99 (1.48)
  Change at Week 7 (n = 103, 97) | -1.98 (2.19) | -1.10 (1.50)
  Change at Week 8 (n = 101, 96) | -1.97 (2.18) | -1.11 (1.59)
  Change at Week 9 (n = 98, 96) | -2.03 (2.13) | -1.11 (1.72)
  Change at Week 10 (n = 97, 90) | -2.18 (2.06) | -1.12 (1.74)
  Change at Week 11 (n = 96, 89) | -2.08 (2.15) | -1.20 (1.85)
  Change at Week 12 (n = 96, 90) | -2.07 (2.21) | -1.20 (1.75)
  Change at Week 13 (n = 93, 90) | -2.08 (2.21) | -1.19 (1.82)
  Change at Week 14 (n = 93, 91) | -2.09 (2.13) | -1.18 (1.83)
  Change at Week 15 (n = 93, 91) | -2.15 (2.10) | -1.11 (1.83)
  Change at Week 16 (n = 89, 89) | -2.25 (2.24) | -1.17 (1.82)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.79, 95% CI 2-sided [-1.23 to -0.35], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week2 A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.87, 95% CI 2-sided [-1.31 to -0.43], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.80, 95% CI 2-sided [-1.24 to -0.36], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.76, 95% CI 2-sided [-1.20 to -0.32], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.94, 95% CI 2-sided [-1.38 to -0.49], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.93, 95% CI 2-sided [-1.37 to -0.48], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 7. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.91, 95% CI 2-sided [-1.35 to -0.47], Standard Error of Mean 0.23
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.90, 95% CI 2-sided [-1.35 to -0.46], Standard Error of Mean 0.23
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Week 9. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.94, 95% CI 2-sided [-1.39 to -0.50], Standard Error of Mean 0.23
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Week 10. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -1.08, 95% CI 2-sided [-1.53 to -0.63], Standard Error of Mean 0.23
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Week 11. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.94, 95% CI 2-sided [-1.39 to -0.49], Standard Error of Mean 0.23
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Week 12. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.92, 95% CI 2-sided [-1.37 to -0.47], Standard Error of Mean 0.23
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Week 13. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.92, 95% CI 2-sided [-1.38 to -0.47], Standard Error of Mean 0.23
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Week 14. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -0.96, 95% CI 2-sided [-1.41 to -0.51], Standard Error of Mean 0.23
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Week 15. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -1.08, 95% CI 2-sided [-1.53 to -0.63], Standard Error of Mean 0.23
Statistical Analysis 16: Comparison: Pregabalin vs Placebo; Week 16. A longitudinal analysis of weekly mean changes using repeated measures mixed models which compared treatments at each week and the last scheduled study week based on this model (to assess durability of treatment effect) was used. Effects for treatment, pooled center, time (week), baseline score, and treatment by time interaction were included as covariates. The covariance structure was compound-symmetric; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significance was declared if p-value <=0.05; LS mean difference = -1.06, 95% CI 2-sided [-1.51 to -0.61], Standard Error of Mean 0.23

9. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory Interference Scale (10-Item) (mBPI-10) Total Score
Description: The Modified Brief Pain Inventory (mBPI-10) Interference Scale is a self administered questionnaire that assessed pain interference with functional activities over the past week. The items were measured on an 11 point scale, ranging from "does not interfere" (0) to "completely interferes" (10). A composite score, the pain interference index, was calculated by averaging the 10 items that comprised the scale.
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline | 4.7 (2.18) | 4.9 (2.21)
  Change from baseline at endpoint (n = 100, 99) | -1.6 (2.19) | -1.1 (2.02)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0438, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline mBPI-10 Total Score as a covariate and pooled center and treatment as fixed (class) cofactors; LS Mean Difference = -0.55, 95% CI 2-sided [-1.08 to -0.02], Standard Error of Mean 0.269

10. Secondary Outcome: Change From Baseline in Quantitative Assessment of Neuropathic Pain (QANeP) - Static Mechanical Allodynia
Description: Participant rated pain scale. The pain produced by the applied stimulus (static mechanical allodynia - gentle constant mechanical pressure) was rated on an 11 point numerical rating scale (0=no pain, 10=worst possible pain).
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 83, 82) | 2.9 (3.16) | 2.6 (2.95)
  Change from baseline at endpoint (n = 79, 75) | -1.0 (2.69) | -0.3 (2.48)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; At/above level: within 2 dermatomes above or below the neurological level of injury (NLI). Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.7103, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline QANeP - Static Mechanical Allodynia as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.17, 95% CI 2-sided [-1.06 to 0.72], Standard Error of Mean 0.448
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Below level: more than 2 dermatomes below the NLI. Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.0747, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 10, analysis 1]; LS mean difference = -0.61, 95% CI 2-sided [-1.28 to 0.06], Standard Error of Mean 0.340

11. Secondary Outcome: Change From Baseline in Quantitative Assessment of Neuropathic Pain (QANeP) - Dynamic Mechanical Allodynia
Description: Participant rated pain scale. The pain produced by the applied stimulus (dynamic mechanical allodynia - gentle stroking with foam brush) was rated on an 11 point numerical rating scale (0=no pain, 10=worst possible pain).
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 83, 82) | 2.7 (2.81) | 2.3 (2.84)
  Change from baseline at endpoint (n = 79, 75) | -0.6 (2.35) | -0.3 (2.32)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; At/Above level Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.5689, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline QANeP - Dynamic Mechanical Allodynia as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.22, 95% CI 2-sided [-0.97 to 0.54], Standard Error of Mean 0.379
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Below level Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.4764, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 11, analysis 1]; LS mean difference = -0.23, 95% CI 2-sided [-0.87 to 0.41], Standard Error of Mean 0.322

12. Secondary Outcome: Change From Baseline in Quantitative Assessment of Neuropathic Pain (QANeP)- Punctata Hyperalgesia
Description: Participant rated pain scale. The pain produced by the applied stimulus (Punctata hyperalgesia - pinprick) was rated on an 11 point numerical rating scale (0=no pain, 10=worst possible pain).
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n=83,82) | 3.9 (3.41) | 3.4 (3.19)
  Change from baseline at endpoint (n=79,75) | -1.0 (2.36) | -0.4 (2.15)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.3362, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline QANeP - Punctate Hyperalgesia as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.46, 95% CI 2-sided [-1.40 to 0.48], Standard Error of Mean 0.474
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.3113, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 12, analysis 1]; LS mean difference = -0.33, 95% CI 2-sided [-0.96 to 0.31], Standard Error of Mean 0.321

13. Secondary Outcome: Change From Baseline in Quantitative Assessment of Neuropathic Pain (QANeP)- Temporal Summation to Tactile Stimuli
Description: Participant rated pain scale. The pain produced by the applied stimulus (Temporal summation to tactile stimuli - repeated touching/tapping) was rated on an 11 point numerical rating scale (0=no pain, 10=worst possible pain).
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 83, 82) | 4.1 (3.54) | 3.9 (3.48)
  Change from baseline at endpoint (n = 79, 75) | -0.5 (2.21) | -0.8 (2.37)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.2721, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline QANeP - Temporal Summation to stimuli as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.60, 95% CI 2-sided [-1.67 to 0.48], Standard Error of Mean 0.539
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.4906, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 13, analysis 1]; LS mean difference = 0.23, 95% CI 2-sided [-0.43 to 0.90], Standard Error of Mean 0.337

14. Secondary Outcome: Change From Baseline in Quantitative Assessment of Neuropathic Pain (QANeP)- Cold Allodynia
Description: Participant rated pain scale. The pain produced by the applied stimulus (Cold allodynia - touch with cool metal rod 13-17 degrees celsius was rated on an 11 point numerical rating scale (0=no pain, 10=worst possible pain).
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 83, 82) | 2.5 (2.97) | 2.7 (3.13)
  Change from baseline at endpoint (n = 79, 72) | -0.1 (2.12) | 0.4 (2.66)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.3123, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline QANeP - Cold Allodynia as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.48, 95% CI 2-sided [-1.42 to 0.46], Standard Error of Mean 0.472
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.1360, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 14, analysis 1]; LS mean difference = -0.55, 95% CI 2-sided [-1.28 to 0.18], Standard Error of Mean 0.368

15. Secondary Outcome: Change From Baseline in Quantitative Assessment of Neuropathic Pain (QANeP)- Cold Hyperalgesia Subscales
Description: Participant rated pain scale. The pain produced by the applied stimulus (Cold hyperalgesia - touch with cold metal rod 4 degrees celsius) was rated on an 11 point numerical rating scale (0=no pain, 10=worst possible pain).
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 83, 82) | 2.8 (3.18) | 2.8 (3.25)
  Change from baseline at endpoint (n = 79, 72) | -0.1 (2.60) | 0.4 (2.82)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.4257, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline QANeP - Cold Hyperalgesia Subscales as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.44, 95% CI 2-sided [-1.53 to 0.65], Standard Error of Mean 0.549
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.2005, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 15, analysis 1]; LS mean difference = -0.53, 95% CI 2-sided [-1.34 to 0.28], Standard Error of Mean 0.412

16. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) - 12 Items Total Intensity Score
Description: Participant rated questionnaire used to evaluate different symptoms of neuropathic pain (dimensions: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia [P/D]). Includes 10 descriptors quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. Questionnaire generates a score in each of the relevant dimensions and a total score of 0-100. Higher score indicates a greater intensity of pain.
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 104, 106) | 0.4 (0.20) | 0.4 (0.22)
  Change from baseline at endpoint (n = 99, 99) | -0.1 (0.21) | -0.1 (0.17)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1377, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline NPSI - 12 Items Total Intensity Score as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.04, 95% CI 2-sided [-0.09 to 0.01], Standard Error of Mean 0.025

17. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) - Burning Spontaneous Pain
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: mITT; LOCF;(n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline | 0.5 (0.32) | 0.5 (0.30)
  Change from baseline at endpoint (n = 100, 99) | -0.1 (0.34) | -0.1 (0.28)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3312, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline NPSI - Burning Spontaneous Pain as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.04, 95% CI 2-sided [-0.11 to 0.04], Standard Error of Mean 0.038

18. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) - Pressing Spontaneous Pain
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline | 0.4 (0.31) | 0.4 (0.31)
  Change from baseline at endpoint (n = 100, 99) | -0.1 (0.28) | -0.0 (0.26)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0440, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline NPSI - Pressing Spontaneous Pain as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.07, 95% CI 2-sided [-0.13 to 0.00], Standard Error of Mean 0.033

19. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) - Paroxysmal Pain
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline | 0.4 (0.29) | 0.3 (0.30)
  Change from baseline at endpoint (n = 100, 99) | -0.1 (0.31) | -0.1 (0.26)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1370, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline NPSI - Paroxysmal Pain as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.05, 95% CI 2-sided [-0.12 to 0.02], Standard Error of Mean 0.033

20. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) - Evoked Pain
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline | 0.4 (0.29) | 0.4 (0.29)
  Change from baseline at endpoint (n = 100, 99) | -0.1 (0.24) | -0.1 (0.22)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8911, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline NPSI - Evoked pain as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = 0.00, 95% CI 2-sided [-0.06 to 0.05], Standard Error of Mean 0.028

21. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) - Paresthesia/Dysesthesia
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 104, 106) | 0.5 (0.28) | 0.5 (0.28)
  Change from baseline at endpoint (n = 99, 99) | -0.1 (0.29) | -0.1 (0.27)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3731, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline NPSI - Paresthesia/Dysesthesia as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.03, 95% CI 2-sided [-0.10 to 0.04], Standard Error of Mean 0.034

22. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) - Individual Item (1, 2, 3, 5, 6, 8, 9, 10, 11, 12) Score
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  1- Burning pain (n = 100, 99) | -1.39 (3.420) | -1.00 (2.825)
  2- Squeezing pain (n = 100, 99) | -1.04 (3.181) | -0.41 (3.110)
  3- Pain like pressure (n = 100, 99) | -0.73 (3.429) | -0.20 (3.326)
  5- Electric shocks (n = 100, 99) | -1.77 (3.426) | -0.68 (3.664)
  6- Stabbing pain (n = 100, 99) | -1.13 (3.541) | -0.52 (2.804)
  8- By light touching (n = 100, 99) | -0.78 (3.080) | -0.94 (2.683)
  9- By pressure (n = 100, 99) | -1.22 (2.784) | -1.10 (2.675)
  10- By something cold (n = 100, 99) | -0.89 (3.372) | -0.52 (2.459)
  11- Pins and needles (n = 99, 99) | -1.01 (3.125) | -0.62 (3.269)
  12- Tingling (n = 99, 99) | -0.99 (3.559) | -0.83 (3.034)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Item 1 - Burning pain Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.3312, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline NPSI - Individual Item Score as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.37, 95% CI 2-sided [-1.13 to 0.38], Standard Error of Mean 0.383
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Item 2 - Squeezing pain Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.0976, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = -0.63, 95% CI 2-sided [-1.37 to 0.12], Standard Error of Mean 0.377
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Item 3 - Pain like pressure Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.0538, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = -0.76, 95% CI 2-sided [-1.54 to 0.01], Standard Error of Mean 0.393
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Item 5 - Electric shocks Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.3239, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = -0.38, 95% CI 2-sided [-1.15 to 0.38], Standard Error of Mean 0.389
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Item 6 - Stabbing pain Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.1912, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = -0.49, 95% CI 2-sided [-1.23 to 0.25], Standard Error of Mean 0.376
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Item 8 - By light touching Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.6720, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = 0.15, 95% CI 2-sided [-0.55 to 0.85], Standard Error of Mean 0.353
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Item 9 - By pressure Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.7821, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = -0.09, 95% CI 2-sided [-0.74 to 0.56], Standard Error of Mean 0.330
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Item 10 - By something cold Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.6851, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = -0.14, 95% CI 2-sided [-0.84 to 0.55], Standard Error of Mean 0.352
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Item 11 - Pins and needles Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.3610, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = -0.35, 95% CI 2-sided [-1.12 to 0.41], Standard Error of Mean 0.387
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Item 12 - Tingling Null hypothesis - the mean of the measure for the pregabalin group was the same as the mean of the measure for the placebo group; Alternative hypothesis - the mean of the measure for the pregabalin group was different from the mean of the measure for the placebo group; Test type: Superiority or Other; p = 0.4915, ANCOVA — Significance was declared if p-value <=0.05; [statistical method as in outcome 22, analysis 1]; LS mean difference = -0.28, 95% CI 2-sided [-1.07 to 0.52], Standard Error of Mean 0.402

23. Secondary Outcome: Number of Participants With Improved Duration of Brief Pain Attacks Based on NPSI - Duration (Item 4)
Description: NPSI - Temporal item which assesses the duration (number of hours during the last 24 hours) of spontaneous ongoing pain. Improved duration would be a decrease in the number of hours of spontaneous ongoing pain during the last 24 hours compared to baseline.
Time Frame: Baseline, Week 16
Population: MITT; LOCF; (N) = number of participants with data available for analysis
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 100 | 97
participants | 39 | 28
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis - The rate of subjects with improvement for the pregabain group was equal to the rate of subjects with improvement for the placebo group; Alternative hypothesis - The rate of subjects with improvement for the pregabain group was not equal to the rate of subjects with improvement for the placebo group; Test type: Superiority or Other; p = 0.0536, Cochran-Mantel-Haenszel — p-values are adjusted for baseline score. Significance was declared if p-value <=0.05

24. Secondary Outcome: Number of Participants With Improvement in the Number of Attacks Based on NPSI - Number of Attacks (Item 7)
Description: NPSI - Temporal item which assesses the paroxysmal pain (number of pain attacks during the last 24 hours). Improvement in the number of attacks would be a decrease in the number of paroxysms during the last 24 hours compared to baseline.
Time Frame: Baseline, Week 16
Population: MITT; LOCF; (N) = number of participants with data available for analysis
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 100 | 99
participants | 48 | 38
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.3107, Cochran-Mantel-Haenszel — p-values are adjusted for baseline score. Significance was declared if p-value <=0.05

25. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS)- 9-Item Overall Sleep Problems Index
Description: Participant rated questionnaire to assess sleep quality and quantity. Consists of a 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); 7 subscales rated 1 (all the time) to 6 (none of the time): sleep disturbance, snoring, awaken short of breath (SOB) or with a headache, somnolence adequacy, and sleep quantity. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range multiplied by 100); total score range = 0 to 100; higher score indicates greater intensity of attribute.
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 105, 103) | 45.7 (18.02) | 45.9 (19.00)
  Change from baseline at endpoint (n = 100, 95) | -10.8 (16.70) | -5.8 (16.21)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0262, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline MOS 9-item Sleep Problems Index as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -4.89, 95% CI 2-sided [-9.19 to -0.59], Standard Error of Mean 2.182

26. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS) - Sleep Disturbance
Description: as for outcome 25
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 105, 104) | 51.9 (25.88) | 51.2 (26.68)
  Change from baseline at endpoint (n = 100, 97) | -17.3 (25.25) | -8.0 (21.70)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0041, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline MOS - Sleep disturbance as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -8.67, 95% CI 2-sided [-14.55 to -2.78], Standard Error of Mean 2.985

27. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS) - Sleep Adequacy
Description: as for outcome 25
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 105, 104) | 42.3 (25.92) | 43.8 (26.92)
  Change from baseline at endpoint (n = 100, 97) | 11.6 (27.26) | 5.7 (28.83)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0998, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline MOS - Sleep Adequacy as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = 5.78, 95% CI 2-sided [-1.11 to 12.66], Standard Error of Mean 3.492

28. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS) - Snoring
Description: as for outcome 25
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 105, 104) | 31.2 (34.07) | 35.6 (35.47)
  Change from baseline at endpoint (n = 100, 97) | 2.2 (25.88) | -4.7 (27.50)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1048, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline MOS - Snoring as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = 5.70, 95% CI 2-sided [-1.20 to 12.61], Standard Error of Mean 3.501

29. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS) - Awaken Short of Breath or With a Headache
Description: as for outcome 25
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 105, 105) | 15.0 (23.00) | 12.8 (23.23)
  Change from baseline at endpoint (n = 100, 98) | -6.2 (22.33) | -0.2 (22.52)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0347, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included baseline MOS - Awaken Short of Breath or with headache as covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -5.14, 95% CI 2-sided [-9.91 to -0.37], Standard Error of Mean 2.417

30. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS) - Sleep Quantity
Description: as for outcome 25
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 104,105) | 5.9 (1.45) | 6.2 (1.64)
  Change from baseline at endpoint (n = 100, 98) | 0.6 (1.42) | 0.2 (1.29)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0436, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline MOS - Sleep Quantity as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = 0.38, 95% CI 2-sided [0.01 to 0.76], Standard Error of Mean 0.189

31. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS) - Somnolence
Description: as for outcome 25
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline (n = 105, 105) | 36.3 (19.81) | 39.7 (23.43)
  Change from baseline at endpoint (n = 100, 97) | -0.8 (20.64) | -4.9 (22.31)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2761, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline MOS - Somnolence as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = 3.02, 95% CI 2-sided [-2.44 to 8.49], Standard Error of Mean 2.770

32. Secondary Outcome: Number of Participants Having Optimal Sleep Based on Medical Outcomes Study Sleep Scale (MOS-SS)
Description: as for outcome 25
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (N) = number of participants with data available for analysis
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 100 | 99
participants | 49 | 30
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis - The rate of subjects with optimal sleep for the pregabain group was equal to the rate of subjects with optimal sleep for the placebo group; Alternative hypothesis - The rate of subjects with optimal sleep for the pregabain group was not equal to the rate of subjects with optimal sleep for the placebo group; Test type: Superiority or Other; p = 0.0024, Regression, Logistic — Significance was declared if p-value <=0.05; Logistic Regression Model included Pooled Center and Treatment as the categorical factors, and Optimal Sleep Score at Baseline as the covariate; Odds Ratio (OR) = 2.81, 95% CI 2-sided [1.443 to 5.491]

33. Secondary Outcome: Change From Baseline in Hospital and Anxiety Depression Scale (HADS) - Anxiety
Description: HADS: participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline | 6.7 (4.41) | 6.9 (4.12)
  Change from baseline at endpoint (n = 100, 99) | -1.4 (3.21) | -0.8 (3.55)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1164, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline HADS - Anxiety as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.68, 95% CI 2-sided [-1.54 to 0.17], Standard Error of Mean 0.433

34. Secondary Outcome: Change From Baseline in Hospital and Anxiety Depression Scale (HADS) - Depression
Description: as for outcome 33
Time Frame: Baseline, Week 16
Population: mITT; LOCF; (n) = number of participants with data available for analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 105 | 106
score on scale
  Baseline | 5.2 (3.96) | 6.3 (3.99)
  Change from baseline at endpoint (n = 100, 99) | -1.0 (3.44) | -0.5 (3.56)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0279, ANCOVA — Significance was declared if p-value <=0.05; ANCOVA model included terms of baseline HADS - Depression as a covariate and pooled center and treatment as fixed (class) cofactors; LS mean difference = -0.99, 95% CI 2-sided [-1.87 to -0.11], Standard Error of Mean 0.447

ADVERSE EVENTS:
Time Frame: Baseline up to and including 28 calendar days after the last administration of the study treatment
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 9/112 | 10/107
Other Adverse Events (participants affected / at risk) | 78/112 | 56/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=112) | Placebo (N=107)
Bradycardia (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood amylase increased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=112) | Placebo (N=107)
Vision blurred (Eye disorders) | 7 | 0
Constipation (Gastrointestinal disorders) | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Dry mouth (Gastrointestinal disorders) | 9 | 3
Nausea (Gastrointestinal disorders) | 6 | 3
Fatigue (General disorders) | 10 | 3
Oedema (General disorders) | 6 | 2
Oedema peripheral (General disorders) | 15 | 5
Pain (General disorders) | 6 | 2
Nasopharyngitis (Infections and infestations) | 13 | 8
Urinary tract infection (Infections and infestations) | 12 | 17
Dizziness (Nervous system disorders) | 22 | 6
Headache (Nervous system disorders) | 8 | 5
Somnolence (Nervous system disorders) | 37 | 14
Insomnia (Psychiatric disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.